CLINICAL TRIAL: NCT05198830
Title: A Phase 2 Randomized Study of the BER Inhibitor TRC102 in Combination With Standard Pemetrexed-Platinum-Radiation in Stage III Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Testing the Addition of an Anti-Cancer Drug, TRC102, to the Usual Chemotherapy Treatment (Pemetrexed, Cisplatin or Carboplatin) During Radiation Therapy for Stage III Non-Squamous Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-14403; NCI-2021-14403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE1522; 10512 (Other: City of Hope Comprehensive Cancer Center LAO); 10512 (Other: CTEP); P30CA043703 (NIH)
Record Dates: First submitted 2022-01-14; First posted 2022-01-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Lung Adenocarcinoma; Lung Large Cell Carcinoma; Lung Non-Squamous Non-Small Cell Carcinoma; Stage III Lung Cancer AJCC v8
MeSH Terms: conditions — Adenocarcinoma of Lung; Lung Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; durvalumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; methoxyamine; Pemetrexed; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (methoxyamine, usual care) (Experimental): Patients receive methoxyamine PO on day 1 of each cycle, pemetrexed IV over 10 minutes on day 1 of each cycle, and cisplatin IV over 60 minutes or carboplatin IV over 30 minutes on day 3 of each cycle. Beginning day 3, patients also undergo radiation therapy daily Monday-Friday. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after cycle 2, patients receive durvalumab IV over 60 minutes every 2 weeks or monthly for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI throughout the trial and FDG-PET/CT scan during screening and optionally on study.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Drug: Methoxyamine; Drug: Pemetrexed; Radiation: Radiation Therapy
- Arm II (usual care) (Active Comparator): Patients receive pemetrexed IV over 10 minutes and cisplatin IV over 60 minutes or carboplatin IV over 30 minutes on day 1 of each cycle. Beginning day 1 of each cycle, patients also undergo radiation therapy daily Monday-Friday. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after cycle 2, patients receive durvalumab IV over 60 minutes every 2 weeks or monthly for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI throughout the trial and FDG-PET/CT scan during screening and optionally on study.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: FDG-Positron Emission Tomography; Procedure: Magnetic Resonance Imaging; Drug: Pemetrexed; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT and FDG-PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI 4736; MEDI-4736; MEDI4736
Procedure: FDG-Positron Emission Tomography — Undergo FDG-PET/CT
  Other Names: FDG; FDG-PET; FDG-PET Imaging
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Methoxyamine — Given PO
  Other Names: TRC102 Base
  Arms: Arm I (methoxyamine, usual care)
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Radiation: Radiation Therapy — Undergo thoracic radiation
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial tests whether TRC102 (methoxyamine hydrochloride) in combination usual care treatment comprised of pemetrexed, cisplatin or carboplatin, and radiation therapy followed by durvalumab works better than the usual care treatment alone to shrink tumors in patients with stage III non-squamous non-small cell lung cancer (NSCLC). TRC102 is in a class of drugs called antineoplastic agents. It blocks the ability of a cell to repair damage to its deoxyribonucleic acid (DNA) and may kill tumor cells. It may also help some anticancer drugs work better. Pemetrexed is in a class of medications called antifolate antineoplastic agents. It works by stopping cells from using folic acid to make DNA and may kill tumor cells. Cisplatin is in a class of medications known as platinum-containing compounds. It works by killing, stopping or slowing the growth of tumor cells. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high energy sources to kill tumor cells and shrink tumors. Giving TRC102 in combination with usual care treatment may be more effective than usual care treatment alone in stabilizing and lengthening survival time in patients with stage III non-squamous NSCLC.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To improve progression-free survival (PFS) from 56% with current standard of care (chemoradiation followed by consolidative durvalumab) to 75% at one year with the proposed combination followed by consolidative durvalumab.

SECONDARY OBJECTIVES:

I. To determine overall survival with the proposed combination therapy. II. To assess the incidence of grade 3 or higher pneumonitis and other toxicities.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive methoxyamine orally (PO) on day 1 of each cycle, pemetrexed intravenously (IV) over 10 minutes on day 1 of each cycle, and cisplatin IV over 60 minutes or carboplatin IV over 30 minutes on day 3 of each cycle. Beginning day 3, patients also undergo radiation therapy daily Monday-Friday. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after cycle 2, patients receive durvalumab IV over 60 minutes every 2 weeks or monthly for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) scan or magnetic resonance imaging (MRI) throughout the trial and fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/CT scan during screening and optionally on study.

ARM II: Patients receive pemetrexed IV over 10 minutes and cisplatin IV over 60 minutes or carboplatin IV over 30 minutes on day 1 of each cycle. Beginning day 1 of each cycle, patients also undergo radiation therapy daily Monday-Friday. Treatment repeats every 21 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Beginning 2-6 weeks after cycle 2, patients receive durvalumab IV over 60 minutes every 2 weeks or monthly for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients also undergo CT scan or MRI throughout the trial and FDG-PET/CT scan during screening and optionally on study.

After completion of study treatment, patients are followed up at 30 days, and then every 3 months for 2 years, followed by every 6 months for an additional 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed adenocarcinoma or large cell carcinoma of the lung with confirmation by immunohistochemistry (histologic tissue diagnosis is preferred, but cytology is acceptable).
* Patients must have newly staged IIIA, IIIB or IIIC disease according to the 8th tumor, node, metastasis (TNM) staging classification and to be considered appropriate candidates for aggressive chemoradiotherapy.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >= 10 mm (>= 1 cm) with CT scan, MRI, or calipers by clinical exam.
* Patients must have diagnosed NSCLC, with no prior overlapping radiation therapy delivered for locally advanced NSCLC. Prior stereotactic radiation therapy for stage I lung cancer without overlapping is allowed. Prior systemic antineoplastic therapy is allowed, as deemed appropriate by the treating physician. Prior surgery is allowed. History of previous stage I NSCLC with new mediastinal nodal recurrence (new stage III are eligible).
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of TRC102 in combination with pemetrexed, cisplatin, and durvalumab in patients < 18 years of age, children are excluded from this study.
* Body weight > 30 kg with acceptable nutritional status based on evaluation by treating physician.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 70%).
* Leukocytes >= 3,000/mcL.
* Hemoglobin >= 9.0 g/dL.
* Absolute neutrophil count >= 1,500/mcL.
* Platelets >= 150,000/mcL.
* Serum bilirubin within normal institutional limits (0 - 1.2 mg/ dl). (This will not apply to patients with confirmed Gilbert's syndrome [persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology], who will be allowed only in consultation with their physician.).
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional upper limit of normal (=< 39 U/L).
* Alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal (=< 52 U/L).
* Creatinine =< 1.3 mg/dL.
* Measured creatinine clearance >= 60 mL/min OR glomerular filtration rate (GFR) >= 50 mL/min/1.73 m^2.
* Acceptable pulmonary function as assessed by treating physician.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  * Women < 60 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).
  * Women >= 60 years of age will be considered post-menopausal.
* Life expectancy >= 12 months.
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen with evidence of at least two undetectable viral loads within the past 6 months on the same regimen; the most recent undetectable viral load must be within the past 12 weeks.
  * They must have a CD4 count of greater than 250 cells/mcL over the past 6 months on this same anti-retroviral regimen and must not have had a CD4 count < 200 cells/mcL over the past 2 years, unless it was deemed related to the cancer and/or chemotherapy induced bone marrow suppression.

    * For patients who have received chemotherapy in the past 6 months, a CD4 count < 250 cells/mcL during chemotherapy is permitted as long as viral loads were undetectable during this same chemotherapy.
  * They must have an undetectable viral load and a CD4 count >= 250 cells/mcL within 7 days of enrollment.
  * They must not be currently receiving prophylactic therapy for an opportunistic infection and must not have had an opportunistic infection within the past 6 months.
  * HIV-infected patients should be monitored every 12 weeks for viral load and CD4 counts.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association functional classification. To be eligible for this trial, patients should be class 2B or better.
* The effects of TRC102 on the developing human fetus are unknown. For this reason and because biochemical inhibitors of the BER pathway agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after completion of durvalumab monotherapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of durvalumab administration, if having sex with women of childbearing potential.
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity who have a legally-authorized representative (LAR) and/or family member available will also be eligible.
* Patients with prior stage I/II non-small cell lung cancer treated with surgery are eligible. Patients with prior stage I NSCLC treated with stereotactic body radiotherapy (SBRT) without overlapping radiation fields would also be eligible. Patients with prior chemotherapy are eligible, at physician's discretion.

Exclusion Criteria:

* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia.
* Patients who are receiving any other investigational agents.
* Patients with treated brain metastases are not eligible as the study is for stage III disease only.
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are not eligible as the study includes only stage III disease.
* Patients with EGFR or ALK mutations are ineligible.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to TRC102 or other agents used in study.
* Patients with uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because TRC102 is a biochemical inhibitor of the BER pathway and durvalumab is an anti-PDL1 antibody, agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with TRC102 or durvalumab, breastfeeding should be discontinued if the mother is treated with TRC102 or durvalumab. These potential risks may also apply to other agents used in this study.

  * Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 6 months after durvalumab monotherapy. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of durvalumab.
* Patients with active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia.
  * Patients with hypothyroidism (e.g. following Hashimoto thyroiditis) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients without active disease in the last 5 years may be included but only after consultation with the study physician.
  * Patients with celiac disease controlled by diet alone.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis [TB] testing in line with local practice), hepatitis B (known positive HBV surface antigen [HBsAg] result), or hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* History of allogenic organ transplantation.
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no active disease before the first dose of investigational product (IP) and of low potential risk for recurrence.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated any carcinoma in situ without evidence of disease.
  * Prostate cancer with stable disease with active or prior treatment that will not interfere with current lung cancer treatment will be eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From randomization to the date of the first documented event of tumor progression or death in the absence of disease progression, assessed at 12 months from randomization and up to 5 years
  PFS primary analysis will be performed using a stratified log-rank test (with the strata being the same as the randomization strata) with a one-sided significance level of 0.10.

SECONDARY OUTCOMES:
Overall survival (OS) | From randomization until death from any cause, assessed up to 5 years
  The analysis of OS will be performed using Kaplan-Meier method with a stratified log-rank test (with the strata being the same as the randomization strata).
Incidence of grade 3 or higher adverse events | Up to 1 year
  Assessed by organ system, by National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Afshin Dowlati, Principal Investigator — Case Western Reserve University
Locations (34):
- United States (34):
  - Keck Medicine of USC Buena Park, Buena Park, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - City of Hope Upland, Upland, California
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Jersey City Medical Center, Jersey City, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm